CLINICAL TRIAL: NCT03735186
Title: Acute Exercise and Coronary Heart Disease Risk Markers in Healthy Male Smokers and Non-Smokers
Brief Title: Exercise and Coronary Heart Disease Risk Markers in Male Smokers and Non-Smokers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Loughborough University (Other)
Collaborators: University of Leicester (Other); University Hospitals, Leicester (Other)
Responsible Party: Principal Investigator, Tareq Alotaibi, Principal investigator, Loughborough University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: R17-P055
Record Dates: First submitted 2018-10-30; First posted 2018-11-08 (Actual); Last update posted 2018-11-09 (Actual); Status verified 2018-11

CONDITIONS: Cigarette Smoking; Coronary Heart Disease; Cardiovascular Risk Factor; Insulin Resistance; Oxidative Stress; Inflammation
Keywords: Coronary heart disease; Exercise; Inflammation; Postprandial lipaemia; Smoking
MeSH Terms: conditions — Cigarette Smoking; Coronary Disease; Insulin Resistance; Inflammation; Motor Activity; Smoking | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Participants will rest in the laboratory on day 1 and day 2 (08:00-17:00). A high fat breakfast and lunch will be consumed on both days at pre-determined intervals.
- Exercise (Experimental): Participants will complete 60 min of treadmill exercise on day 1 (14:30-15:30). Participants will rest in the laboratory for the remainder of day 1 and throughout day 2 (08:00-17:00). A high fat breakfast and lunch will be consumed on both days at pre-determined intervals.
  Interventions: Behavioral: Exercise

INTERVENTIONS:
Behavioral: Exercise — 60 min treadmill exercise performed at 60% of maximum oxygen uptake.
  Arms: Exercise

SUMMARY:
The present study will investigate the effect of acute exercise on fasting and postprandial risk markers for coronary heart disease (CHD) in healthy male cigarette smokers and non-smokers.

Participants will complete two, 2-day trials in a random crossover design separated by an interval of at least 1 week. On day 1, participants will rest (control) or complete 60 minute of treadmill exercise at 60% of maximum oxygen uptake (exercise). On day 2, participants will rest and consume two high fat meals (breakfast and lunch) over an 8-h period during which 13 venous blood samples and nine blood pressure measurements will be taken at pre-determined intervals.

It is hypothesised that men who smoke cigarettes will exhibit impaired fasting and postprandial metabolic risk markers compared to non-smokers, but a single bout of exercise will be equally, if not more, efficacious for improving the CHD risk factor profile in smokers than non-smokers.

DETAILED DESCRIPTION:
Cigarette smoking is a strong and independent risk factor for CHD and is associated with impaired postprandial metabolism. Previous studies suggest that postprandial metabolism and other risk markers for CHD can be improved with acute exercise in healthy non-smokers, but less is known about responses in cigarette smokers. Therefore, the present study will compare the effect of acute exercise on fasting and postprandial risk markers for CHD in healthy male cigarette smokers and non-smokers.

A total of 12 healthy male cigarette smokers and 12 healthy male non-smokers matched for age and body mass index will be recruited. Before the main experimental trials, participants will attend the laboratory for a preliminary visit to complete screening questionnaires and to undergo familiarisation, anthropometric measurements (stature, body mass, waist and hip circumference, body fat) and exercise testing to determine maximum oxygen uptake.

Participants will complete two, 2-day (08:00-17:00) experimental trials in a randomised cross over design: control and exercise. On day 1, participants will arrive at the laboratory at 08:00 having fasted overnight and a baseline fasting venous blood sample and blood pressure measurement will be taken. A high fat breakfast and lunch meal will be consumed at 08:30 and 12:00, respectively. The control and exercise trials will be identical, except a 60 min bout of treadmill exercise at 60% of maximum oxygen uptake will be performed at 14:30 in the exercise trial.

On day 2, participants will arrive at 08:00 having fasted overnight for 10 h and will rest in the laboratory until 17:00. Participants in the smokers group will be asked to stop smoking at 08:00. A high fat breakfast and lunch will be consumed at 09:00 and 13:00, respectively. Venous blood samples from a cannula will be collected in the fasted state and at 0.25, 0.5, 1, 2, 3, 4, 4.25, 4.5, 5, 6, 7 and 8 h after the breakfast meal. Resting arterial blood pressure will be measured in the fasted state and at hourly intervals thereafter.

ELIGIBILITY:
Inclusion criteria:

* 20- to 45-year-old healthy male smokers or non-smokers;
* Be able to exercise continuously for 1 hour;
* Body mass index between 18.5 and 29.9 kg/m2;
* Weight stable for the past 3 months;
* No known contradictions to maximal exertion exercise (e.g., recent musculoskeletal injury, congenital heart disease).
* A regular cigarette smoker or non-smoker for the last 12 months according to the definition below;

The National Health Interview Survey (NHIS) definitions will be used to identify cigarette smokers and non-smokers (Link: NHIS Adult Tobacco Use):

1. Current smokers will be defined as an adult who has smoked ≥100 cigarettes in their lifetime and who currently smokes cigarettes every day.
2. Non-smokers will be defined as an adult who has never smoked or who has smoked < 100 cigarettes in their lifetime

The following questions will determine the eligibility and group allocation:

1. Do you currently smoke cigarettes on a daily basis?
2. Have you smoked at least 100 cigarettes in your entire life?

If the person answers YES to Q1 and YES to Q2 they are eligible for the study and will be allocated to the smokers group.

If the person answers NO to Q1 and NO to Q2 they are eligible for the study and will be allocated to the non-smokers group.

Individuals answering any other combination (YES, NO or NO, YES) will not be eligible to take part in the study.

Exclusion Criteria:

* Not meeting the criteria for a smoker or non-smoker (defined above);
* Current E-Cigarette smoker;
* Musculoskeletal injury that has affected normal ambulation within the last month;
* Any muscle or bone injuries that do not allow them to walk and run on a treadmill;
* Uncontrolled exercise-induced asthma;
* Heart conditions;
* Coagulation or bleeding disorders;
* Diabetes (metabolism will be different to non-diabetics potentially skewing the data);
* Taking any medication that might influence fat metabolism;
* Taking any medication that might influence blood glucose (e.g., insulin for diabetes);
* Dieting or restrained eating behaviours;
* Weight fluctuation greater than 3 kg in the 3 months prior to study enrolment;
* A food allergy.

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2017-08-04 (Actual); Primary Completion 2018-10-02 (Actual); Study Completion 2018-10-02 (Actual)

PRIMARY OUTCOMES:
Triacylglycerol concentration | 8 hours (Plasma samples will be collected at 0 (fasted), 0.25, 0.5, 1, 2, 3, 4, 4.25, 4.5, 5, 6, 7, 8 hours)
  Total area under the plasma triacylglycerol concentration versus time curve on day 2

SECONDARY OUTCOMES:
Glucose concentration | 8 hours (Plasma samples will be collected at 0 (fasted), 0.25, 0.5, 1, 2, 3, 4, 4.25, 4.5, 5, 6, 7, 8 hours)
  Time-course of plasma glucose concentrations on day 2 of the exercise and control trials.
Insulin concentration | 8 hours (Plasma samples will be collected at 0 (fasted), 0.5, 1, 3, 4, 4.5, 6, 8 hours)
  Time-course of plasma insulin concentrations on day 2 of the exercise and control trials.
Homeostasis model assessment of insulin resistance (HOMA-IR) | Fasting (Plasma samples will be collected at 0 (fasted) hours)
  Homeostasis model assessment of insulin resistance (HOMA-IR) on day 2 of the exercise and control trials using fasting glucose and insulin concentrations.
Non-esterified fatty acids concentration | 8 hours (Plasma samples will be collected at 0 (fasted), 0.5, 1, 3, 4, 4.5, 6, 8 hours)
  Time-course of plasma non-esterified fatty acid concentrations on day 2 of the exercise and control trials.
Total cholesterol concentration | Fasting (Plasma samples will be collected at 0 (fasted) hours)
  Circulating concentrations of plasma total cholesterol in the fasted state on day 2 of the exercise and control trials.
High-density lipoprotein cholesterol concentration | Fasting (Plasma samples will be collected at 0 (fasted) hours)
  Circulating concentrations of plasma high-density lipoprotein cholesterol in the fasted state on day 2 of the exercise and control trials.
Low-density lipoprotein cholesterol concentration | Fasting (Plasma samples will be collected at 0 (fasted) hours)
  Circulating concentrations of plasma low-density lipoprotein cholesterol in the fasted state on day 2 of the exercise and control trials.
C-reactive protein concentration | 8 hours (Plasma samples will be collected at 0 (fasted), 2, 5, 8 hours)
  Time-course of plasma C-reactive protein concentrations on day 2 of the exercise and control trials.
Interleukin-6 concentration | 8 hours (Plasma samples will be collected at 0 (fasted), 2, 5, 8 hours)
  Time-course of plasma interleukin-6 concentrations on day 2 of the exercise and control trials.
Interleukin-10 concentration | 8 hours (Plasma samples will be collected at 0 (fasted), 2, 5, 8 hours)
  Time-course of plasma interleukin-10 concentrations on day 2 of the exercise and control trials.
Tumor necrosis factor alpha concentration | 8 hours (Plasma samples will be collected at 0 (fasted), 2, 5, 8 hours)
  Time-course of plasma tumor necrosis factor alpha concentrations on day 2 of the exercise and control trials.
Peroxiredoxin-4 concentration | 8 hours (Plasma samples will be collected at 0 (fasted), 2, 5, 8 hours)
  Time-course of plasma peroxiredoxin-4 concentrations on day 2 of the exercise and control trials.
Superoxide dismutase 3 concentration | 8 hours (Plasma samples will be collected at 0 (fasted), 2, 5, 8 hours)
  Time-course of plasma superoxide dismutase 3 concentrations on day 2 of the exercise and control trials.
Systolic and diastolic blood pressure | 8 hours (Blood pressure will be measured at 0 (fasted), 1, 2, 3, 4, 5, 6, 7, 8 hours)
  Time-course of systolic and diastolic blood pressure on day 2 of the exercise and control trials.

CONTACTS AND LOCATIONS:
Overall Officials: David Stensel, Principal Investigator — Loughborough University; Tareq Alotaibi, Principal Investigator — Loughborough University
Locations (1):
- Loughborough University, Loughborough, Leicestershire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Arjunan SP, Deighton K, Bishop NC, King J, Reischak-Oliveira A, Rogan A, Sedgwick M, Thackray AE, Webb D, Stensel DJ. The effect of prior walking on coronary heart disease risk markers in South Asian and European men. Eur J Appl Physiol. 2015 Dec;115(12):2641-51. doi: 10.1007/s00421-015-3269-7. Epub 2015 Oct 5. PMID 26438068
- [Background] Arjunan SP, Bishop NC, Reischak-Oliveira A, Stensel DJ. Exercise and coronary heart disease risk markers in South Asian and European men. Med Sci Sports Exerc. 2013 Jul;45(7):1261-8. doi: 10.1249/MSS.0b013e3182853ecf. PMID 23470315
- [Background] Miyashita M, Burns SF, Stensel DJ. Accumulating short bouts of brisk walking reduces postprandial plasma triacylglycerol concentrations and resting blood pressure in healthy young men. Am J Clin Nutr. 2008 Nov;88(5):1225-31. doi: 10.3945/ajcn.2008.26493. PMID 18996856
- [Derived] Alotaibi TF, Thackray AE, Roberts MJ, Alanazi TM, Bishop NC, Wadley AJ, King JA, O'Donnell E, Steiner MC, Singh SJ, Stensel DJ. Acute Running and Coronary Heart Disease Risk Markers in Male Cigarette Smokers and Nonsmokers: A Randomized Crossover Trial. Med Sci Sports Exerc. 2021 May 1;53(5):1021-1032. doi: 10.1249/MSS.0000000000002560. PMID 33196606

DOCUMENTS (1):
  • Statistical Analysis Plan (2018-10-23): https://cdn.clinicaltrials.gov/large-docs/86/NCT03735186/SAP_001.pdf